CLINICAL TRIAL: NCT03221153
Title: Simulation for the Evaluation of General Skills in Patient Safety and Quality in Undergraduate Medical Students
Brief Title: Patient Safety Skills for Medical Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Tecnologico y de Estudios Superiores de Monterey (Other)
Responsible Party: Principal Investigator, Karla Patricia Pacheco Alvarado, MD, Instituto Tecnologico y de Estudios Superiores de Monterey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EGSPQS
Record Dates: First submitted 2016-07-29; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: Patient Safety; Quality; Simulation; Undergraduate; Medical Student
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial of two educational interventions
Who Masked: Outcomes Assessor
Masking Description: Masking only at the level of outcome assessor as this is an educational intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (No Intervention): This is the control group. Participants in this group will take the usual course without simulation techniques.
- Simulation (Experimental): This is the intervention group. Participants in this group will to take the course with simulation techniques.
  Interventions: Procedure: Simulation techique

INTERVENTIONS:
Procedure: Simulation techique — The intervention group will be in a simulated case with mock scenarios and interaction by 'acting out' the clinical situation where knowledge and attitudes about safety in hospitalized patients will be assessed.
  Arms: Simulation

SUMMARY:
In this project, the authors aim to evaluate the use of high fidelity simulation as a method of evaluation of general skills in fifth year medical students about patient quality and safety in a hospital setting.

DETAILED DESCRIPTION:
Undergraduate training in patient safety and healthcare quality is often overlooked by medical curricula.

Simulation techniques have been used in different subjects as a support for learning invasive techniques in surgical areas, but it has not been used to improve knowledge and performance on patient quality domains that would be applied in real life scenarios.

This project is a randomized trial for medical students undertaking the course in "Quality and Patient Safety". The authors will randomized students at the beginning of each rotation into two groups: a) an intervention group (where students will take the simulation and will be evaluated by a final written exam); and b) a control group (where students will take only the usual teaching in classrooms and will be evaluated with the same written exam). Furthermore, students will be asked to fill a questionnaire to obtain their attitudes and knowledge about the topics in quality and safety in healthcare.

ELIGIBILITY:
Inclusion Criteria:

* 5th year medical students enrolled in the course "Quality and Patient Safety" in the Tecnológico de Monterrey School of Medicine, Campus Monterrey.

Ages: 21 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-08-25; Primary Completion 2017-09-01 (Estimated); Study Completion 2017-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean score of skills and knowledge about quality and patient safety | One year
  Assessed by questionnaire evaluation of knowledge in the area of patient safety and quality of healthcare using a multiple choice question examination and a survey. This outcome is measured in a scale from 0 to 100 individually and it will be averaged throughout each group.

SECONDARY OUTCOMES:
Qualitative Evaluation of Attitudes and preferences towards patient safety | One year
  Assessed by interview of individuals about their attitudes and behaviours

CONTACTS AND LOCATIONS:
Overall Officials: Karla Pacheco, MD, Principal Investigator — Instituto Tecnologico y de Estudios Superiores de Monterey
Locations (1):
- Tecnologico de Monterrey School of Medicine, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Miller GE. The assessment of clinical skills/competence/performance. Acad Med. 1990 Sep;65(9 Suppl):S63-7. doi: 10.1097/00001888-199009000-00045. No abstract available. PMID 2400509
- [Result] Sperling JD, Clark S, Kang Y. Teaching medical students a clinical approach to altered mental status: simulation enhances traditional curriculum. Med Educ Online. 2013 Apr 3;18:1-8. doi: 10.3402/meo.v18i0.19775. PMID 23561054